CLINICAL TRIAL: NCT01245036
Title: Rifampicin and Isoniazid Along With Prednisolone Compared to Prednisolone Alone in Treatment of Sarcoidosis: a Pilot Randomized Controlled Trial
Brief Title: Efficacy of Antituberculous Therapy in Management of Sarcoidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sarc/Att/01
Record Dates: First submitted 2010-11-15; First posted 2010-11-22 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Sarcoidosis; Tuberculosis
Keywords: Sarcoidosis; Tuberculosis
MeSH Terms: conditions — Sarcoidosis; Tuberculosis | interventions — Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Glucocorticoid arm (Active Comparator): Prednisolone 0.75 mg/kg/day for 6 weeks (maximum 60 mg) Prednisolone 0.5 mg/kg/day for 6 weeks (maximum 40 mg) Prednisolone 0.25 mg/kg/day for 6 months (maximum 20 mg) Taper over the next three months Prednisolone 0.25 mg/kg EOD for 15 days Prednisolone 0.125 mg/kg EOD for 15 days Then taper by 5 mg every 15 days to complete one year
  Interventions: Drug: Antituberculous therapy along with steroids

INTERVENTIONS:
Drug: Antituberculous therapy along with steroids — INH (300 mg/day) plus Rifampicin (450 mg/day if wt.<50 kg and 600 mg/day if wt. >50 kg) for six months Prednisolone 1 mg/kg/day for 6 weeks (maximum 80 mg) Prednisolone 0.75 mg/kg/day for 6 weeks (maximum 60 mg) Prednisolone 0.5 mg/kg/day for 3 months (maximum 40 mg) Prednisolone 0.25 mg/kg/day for 3 months (maximum 20 mg) Taper over the next three months Prednisolone 0.25 mg/kg EOD for 15 days Prednisolone 0.125 mg/kg EOD for 15 days Then taper by 5 mg every 15 days to complete one year

SUMMARY:
From the time sarcoidosis has been described, there has always been a belief that the disease is in some way related to tuberculosis. If indeed tuberculosis is a causal factor in sarcoidosis, then the hypothesis can be further reinforced, if anti-tubercular therapy (ATT) is useful in treatment of sarcoidosis. Very few trials have been conducted in the past but the results of these trials have been discouraging. These trials were generally small studies and limited by time bias and used older regimens based on isoniazid, amino-salicylic acid and streptomycin. In our experience nearly one third of patients who are finally diagnosed to have sarcoidosis, have received ATT for variable length of time, but its impact of final outcome of sarcoidosis has not been studied. The aim of this prospective randomized controlled trial (RCT) is to evaluate the efficacy and safety of Rifampicin and Isoniazid along with prednisolone compared to prednisolone alone in treatment of Sarcoidosis.

DETAILED DESCRIPTION:
Sarcoidosis has evolved from the position of a disease of relative obscurity in the tropics, towards an increasing recognition and reporting from India and around. From the time sarcoidosis has been described, there has always been a belief that the disease is in some way related to tuberculosis. However, the inability to identify mycobacteria by histologic staining or culture from pathologic tissues continues to be one of the strongest arguments against a potential role for mycobacteria. Of late, molecular analysis (such as polymerase chain reaction [PCR] techniques) for nucleic acids of the putative agents serves as an alternative method for isolating fastidious organisms. A recent meta-analysis suggested a 30% prevalence rate of mycobacterial DNA in sarcoid samples but the individual studies reported detection rates from 0-50%. Moreover, most of these studies were published from countries with low prevalence for tuberculosis. If indeed mycobacteria are etiologically linked to sarcoidosis then the detection rates for mycobacterial DNA in sarcoid samples would be higher in countries with high prevalence of TB. In a recent prospective case-control study aimed at detection of mycobacterial DNA in patients with sarcoidosis from India, reinforced the hypothesis by showing mycobacterial DNA with PCR for 65 kDa protein gene in 48% of samples (BAL or biopsy) from freshly diagnosed patients of sarcoidosis.

There are numerous factors that favor mycobacteria being a trigger for sarcoidosis. These include histopathological appearances of the granulomas 15, reports of mycobacterial disease either existing coincidentally, succeeding or antedating sarcoidosis and the finding of mycobacteria in occasional granulomas of sarcoidosis.Passage experiments have also suggested that mycobacteria with characteristics of M. tuberculosis may be the incriminating agent.Recent studies on humoral immunity to mycobacterial antigens from sarcoidosis patients have renewed interest in a potential of mycobacteria in sarcoidosis. It has been shown that mycobacterial ESAT-6 and katG are recognized by sarcoidosis CD4+ T cells when presented by known sarcoidosis susceptibility allele, DRB1*1101. It is possible that the presence of mycobacterial infection or BCG vaccination in genetically predisposed host may be involved in the development of autoimmunity.It has also been suggested that the organism might exist in a cell wall deficient L-form and may be difficult to isolate.

This possible link not only has implications in the differential diagnosis of the two common conditions, it may also have some therapeutic implications. Reactivation of tuberculosis after cortico-steroid treatment is instituted for sarcoidosis is a genuine concern, given the high prevalence of latent infection in our country. If indeed tuberculosis is a causal factor in sarcoidosis, then the hypothesis can be further reinforced, if anti-tubercular therapy (ATT) is useful in treatment of sarcoidosis. Very few trials have been conducted in the past but the results of these trials have been discouraging. These trials were generally small studies and limited by time bias and used older regimens based on isoniazid, amino-salicylic acid and streptomycin. In our experience nearly one third of patients who are finally diagnosed to have sarcoidosis, have received ATT for variable length of time, but its impact of final outcome of sarcoidosis has not been studied.

The aim of this prospective randomized controlled trial (RCT) is to evaluate the efficacy and safety of Rifampicin and Isoniazid along with prednisolone compared to prednisolone alone in treatment of Sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

newly diagnosed sarcoidosis defined by presence of all of the following criteria:

1. Presence with clinical features of pulmonary (dyspnea, dry cough, chest pain, fever, fatigue or crackles) or extra pulmonary organ (lymph nodes, liver, spleen, skin, eyes, heart, etc.) involvement and consistent radiological involvement and
2. Compact non-caseating granulomas on trans-bronchial biopsy which are tissue AFB smear-negative

Exclusion Criteria:

Patients who have received glucocorticoid treatment before initial evaluation by us, or with presence of concomitant other cardio pulmonary disease will be excluded.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Remission rates | Three months

SECONDARY OUTCOMES:
Relapse rates in the two groups | six and 12 months after completion of treatment
Treatment related adverse effects in the two groups. | Through out

CONTACTS AND LOCATIONS:
Overall Officials: Dheeraj Gupta, Principal Investigator — PGIMER, Chandigarh
Locations (1):
- Deaprtment of Pulmonary Medicine, PGIMER, Chandigarh, Chandigarh, India